CLINICAL TRIAL: NCT04230096
Title: Effect Of Low Level Laser Therapy on Tooth Movement,Gingival,Periodontal Tissue And Pain In Fixed Orthodontic Treatment
Brief Title: Effects Of Low Level Laser Therapy On Tooth Movement,Treatment Related Complications Of Gingivitis,Periodontitis And Pain In Fixed Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, kishore kumar, Consultant, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: kishore kumar
Record Dates: First submitted 2019-12-02; First posted 2020-01-18 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Gingivitis; Pain; Periodontitis; Tooth Migration
Keywords: pain; complications; movement; orthodontic; duration
MeSH Terms: conditions — Gingivitis; Pain; Periodontitis; Tooth Migration | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: This will be an experimental; case controlled study
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- applied group (Experimental): low level laser therapy applied in one group
  Interventions: Device: low level laser therapy
- controlled group (No Intervention): other group will be controlled in which low level laser will not be applied

INTERVENTIONS:
Device: low level laser therapy — apply low level laser therapy on buccal surface of maxillary jaw on anterior segment for three minutes at every three weeks in fixed orthodontic patients in their regular follow up visits
  Other Names: LLLT
  Arms: applied group

SUMMARY:
INTRODUCTION Orthodontic treatment objectives are achieved through the movement of teeth with the application of an external physical force. It takes around 2 to 3 years to finish the treatment.The most common complications associated with orthodontic treatment are

1. Pain
2. Prolonged duration
3. Gingival and Periodontal complications So orthodontists, clinicians and researchers are always looking for some non-invasive and reliable techniques to minimize the possibility of occurrence of these complications.

General objective The prime aim of this research is to study the effect of LLLT on tooth movement,pain, gingival and periodontal complications associated with tooth movement in initial phase of orthodontic treatment.

Design of study This will be an experimental; case controlled study utilizing Low Level Laser Therapy in arch form of application.Anterior teeth segment of the maxillary jaw will be treated with LLLT in one group and other group of patients considered as control.

Study population and samples This research will be conducted among Pakistani subjects who will be going for fix orthodontic treatment. Research subjects will be gathered from Aga Khan Hospital for Women Karimabad A secondary hospital of Aga Khan University Hospital of Karachi Pakistan. The duration of the study will be six months in which each patient will avail their regular follow up orthodontic treatment visits at every three weeks LLLT will be applied at every visit i.e. 0, 1, 2, 3, 4, 5 and 6th visits on anterior segment of the maxillary jaw in one group of patients, while the other group of patients will be controlled.

The clinical parameters gingival index (GI), Bleeding on Probing (BOP), Probing Depth (PD) and clinical attachment loss (CAL) for the research will be recorded at 0, first, third and sixth visit. Study models to determine tooth movement will be taken in all visits from 0 to 6th visit.

A Per forma to record the level of pain has been designed which will be given to all the patients at 0 to sixth all visits to record the pain intensity. Data will be recorded simultaneously.

Sample frame The sample frame of patient recruitment for this research will be consisting of patients who will sign consent for this research and fulfill the inclusion and exclusion criteria. Sample size will be comprised of 88 pre-orthodontic patients, with an age range of 18 to 30 years.

Sample size calculation Sample size will be determined by using PS software (version 3.1.2). To avoid individual variations, the patients will be divided into two groups randomly, using computer generated random numbers. Microsoft Excel 2013 will be used for group randomization. Group A and B will comprise of 36 patients (18 males and 18 females in each group) respectively and only Group A will receive LLLT on anterior segment of the maxillary jaw. However 20% drop out is considered which makes the sample size of 44 in each group at the beginning of study.

Research tool The duration of the study will be 6 months in which each patient will visit on their regular follow up orthodontic treatment visits at every 3 weeks. LLLT will be applied at every visit i.e. 0, 1, 2, 3, 4, 5 and 6 months in patients of Group A. The clinical parameters Gingival Index, Bleeding on Probing (BOP), Probing Depth (PD) and Clinical Attachment Loss (CAL) for the research will be as recorded at 0, first, third and sixth visit of all patients of both groups.

Conclusion The benefits of adopting LLLT (Low Level Laser Therapy) in an arch form in a routine orthodontic practice may enhance the rate of tooth movement, may be helpful to control orthodontic treatment related complications like pain, gingivitis and periodontitis with comfort and without disturbing patient regular recall visits.

DETAILED DESCRIPTION:
INTRODUCTION Background Orthodontic treatment should be based on potential risks and benefit ,pledges appropriate positioning of teeth, corrects jaws and occlusal relationship that enhances mastication, speech, facial aesthetics and also promotes oral and general health which in its turn improves self-confidence of patient, thus bettering quality of life.

Orthodontic treatment objectives are achieved through the movement of teeth with the application of an external physical force. It takes around 2 to 3 years to finish the treatment. However, long duration of treatment and presence of orthodontic appliances is also associated with some risks and complications.

For above mentioned reasons, orthodontists and clinicians have been searching for effective methods to reduce patient discomfort, pain, longest duration of treatment and overcome treatment related gingival and periodontal issues that are not associated with undesirable effects over the course of treatment and on patient health.

For several years, research in laser endorses its use in the treatments involving clinical dentistry and is progressing gradually. Many practitioners have an association of love/hate relationship with bleaching lights and lasers. Laser phototherapy is non- invasive, non- pharmacological, has very rare adverse effects, is pain free and adores a high acceptance from clinicians and also patients.

Justification of the study orthodontic treatment is associated with some complications, particularly its long duration of treatment, and possibility of some adverse effects of treatment like pain, gingivitis and periodontitis, which are extremely bothersome for patients as well as practitioners.The use of LLLT is promising due to it's a non-invasive technique and has been reported with positive results for orthodontic tooth movements, pain and also in cases of gingival and periodontal complications by a number of previous studies.

Previous all studies were done by applying laser on different points through fiber optic tip that is a time-consuming procedure but never, ever arch form of laser has been used so for in the field of orthodontics.

The benefits of adopting LLLT (Low Level Laser Therapy) in an arch form in a routine orthodontic practice may enhance the rate of tooth movement, may be helpful to control orthodontic treatment related complications like pain, gingivitis and periodontitis with comfort and without disturbing patient regular recall visits.

Objectives of the study General objective The prime aim of this research is to study the effect of LLLT on orthodontic patient management. Patient management includes the tooth movement acceleration, pain, gingival and periodontal complications associated with tooth movement in initial phase of orthodontic treatment.

Specific objectives To compare the effect of LLLT on tooth movement applied group and control group with conventional brackets system.

To compare the effect of LLLT on the reduction of pain on applied group and control group with conventional brackets.

To compare the effect of LLLT on applied group and control group on Gingival Index with conventional brackets.

To compare the effect of LLLT on applied group and control group on the Bleeding on Probing (BOP) with conventional brackets To compare the effect of LLLT on applied group and control group on Probing Depth (PD) with conventional brackets.

To compare the effect of LLLT on applied group and control group on clinical attachment loss (CAL) with conventional brackets.

MATERIALS AND METHODS Ethical approval Ethical approval has been obtained from the Human Research and Ethics Committee (HREC), Universiti Sains Malaysia and will be in process from the ethical review committee of the Aga Khan University Hospital of Karachi Pakistan Design of study This will be an experimental; case controlled study utilizing Low Level Laser Therapy in arch form of application to check tooth movement, treatment related pain, gingival and periodontal condition during initial stage of orthodontic treatment. Anterior teeth segment of the maxillary jaw will be treated with LLLT in one group and other group of patients considered as control.

Study population and samples This research will be conducted among Pakistani subjects who will be going for fix orthodontic treatment. Research subjects will be gathered from Aga Khan Hospital for Women Karimabad A secondary hospital of Aga Khan University Hospital of Karachi Pakistan. The duration of the study will be six months in which each patient will avail their regular follow up orthodontic treatment visits at every three weeks and further required orthodontic treatment will be continue under supervision of principal investigator and field supervisor.

LLLT will be applied at every visit i.e. 0, 1, 2, 3, 4, 5 and 6th visits on anterior segment of the maxillary jaw in one group of patients, while the other group of patients will be controlled.

The procedure will be performed in an isolated room, using protective eye-wear for the patient, operator and dental assistant because the unprotected human eye is extremely sensitive to laser radiation due to tissue characteristics.

The clinical parameters gingival index (GI), Bleeding on Probing (BOP), Probing Depth (PD) and clinical attachment loss (CAL) for the research will be recorded at 0, first, third and sixth visit.

Study models to determine tooth movement will be taken in all visits from 0 to 6th visit.

A Performa to record the level of pain has been designed which will be given to all the patients at 0 to sixth all visits to record the pain intensity. Data will be recorded simultaneously.

Sample frame The sample frame of patient recruitment for this research will be consisting of patients who will sign consent for this research and fulfill the inclusion and exclusion criteria. Our sample will be comprised of 88 pre-orthodontic patients, with an age range of 18 to 30 years.

Inclusion criteria

1. Selected patients will be Pakistani in origin.
2. Age 18 to 30 years.
3. Patients with class 1 with mild crowding.
4. Patient with healthy periodontium.
5. Patients who will about to get their fixed orthodontic treatment started with the conventional ligated brackets.
6. Patients who will sign consent for participation in research and use of collected specimen/data for future reference.
7. Patients with ovoid arch form to compact with laser assisted tray. Exclusion criteria Patients on medications which alter the gingival health e.g. Phenytoin (Dilantin), Cyclosporine A (Sandimmun), Nifedipine (Adalat), Corticosteroids, contraceptive pills.

Patients on those medications which alter the bone metabolism or tooth movement e.g. NSAIDs, Corticosteroids, Bisphosphonates etc.

Patients with following disorder: Diabetes Type 1 and 2, Osteoporosis, Platelet disorders, Vitamin C deficiency, vascular conditions, Leukemia, HIV infection, crohn's disease.

Patients with pregnancy. Patients with para functional habits, TMJ dysfunction, craniofacial malformation, multiple missing teeth, impacted teeth except third molars, or periodontal compromised patients will be excluded from the study.

Sample Size Calculation Sample size will be determined by using PS software (version 3.1.2). Sample size calculation is based on the specific objective related to the effect of LLLT on tooth movement, treatment induced pain GI, BOP,CAL and PD in initial phase of orthodontic treatment and considering 1 mm mean difference as clinically meaningful .

To avoid individual variations, the patients will be divided into two groups randomly, using computer generated random numbers. Microsoft Excel 2013 will be used for group randomization. Group A and B will comprise of 36 patients (18 males and 18 females in each group) respectively and only Group A will receive LLLT on anterior segment of the maxillary jaw. However 20% drop out is considered which makes the sample size of 44 in each group at the beginning of study.

Research tool Alignment and leveling will be initiated with 0.014-in heat-activated nickel-titanium (NiTi) wire, and later sequences of wires will be 0.016-in NiTi, 0.017 x 0.025-in NiTi, (SS), and 19 X 25-in NiTi. After completion of first stage a final working wire of 0.019 x 0.025 SS will be placed for alignment and leveling.

Application of LLLT will be started on the same day of appliance of brackets according to the group randomization. Procedure will be repeated after every 3 weeks on their regular follow up visits.

Alginate impressions will be made before beginning of retraction (T0) and then will be repeated at every visit till T6. Dental casts will be scanned with micro CT scanner for the analyses explained in the section later.

The duration of the study will be 6 months in which each patient will visit on their regular follow up orthodontic treatment visits at every 3 weeks. LLLT will be applied at every visit i.e. 0, 1, 2, 3, 4, 5 and 6 months in patients of Group A.

The clinical parameters Gingival Index, Bleeding on Probing (BOP), Probing Depth (PD) and Clinical Attachment Loss (CAL) for the research will be as recorded at 0, first, third and sixth visit of all patients of both groups. Data will be recorded simultaneously and will be kept safely for future reference because the treatment of participants will be continued for next more than one year after completion of this study.

Laser specification Gallium-Aluminium-Arsenide (Ga-Al-As) diode laser (Lasotronix, Poland) with a wavelength at 635 nm /200 mW in a continuous (CW) mode of operation will be used.

A Laser assisted teeth whitening trays of 3 cm 2 diameter deliver the laser beam. Irradiation will be performed keeping laser assisted whitening tray in direct contact with the mucosa.

Laser assisted whitening tray will be applied on only buccal side of anterior segment of maxilla in experimental group of patients. 200mW laser output power will be selected. Since the irradiation will be performed for 3 min on anterior segment of maxillary jaw, this makes total energy of 12.5 Joules per session.

Energy density = laser output power x sec / diameter in cm2 To avoid individual variations, randomized controlled trial (RCT) design will be used assigning experimental group and control group randomly. All the patients of Group A will received LLLT on their regular orthodontic visits at three weeks intervals and other patients of Group B will be control.

To test intra-examiner reliability for index reproducibility the examiner will perform duplicate examinations on four subjects using the gingival index (GI), bleeding on probing (BOP), probing depth (PD) and clinical attachment loss (CAL).

To test intra-examiner reliability for index reproducibility the examiner performed duplicate examinations on five subjects using the plaque index (PI), gingival index (GI), gingival bleeding index system (GBI) and pocket probing depth. The test showed very good intra-examiner repeat ability.

Analyses and Measurements:

Gingival index (GI) Introduced by Loe and Silness in 1963, the examination was performed by using a blunt probe.

Score Criteria No inflammation Mild inflammation, slight change in color, slight edema, no bleeding on probing (Mild Gingivitis) Moderate inflammation, moderate glazing, redness, bleeding on probing (Moderate Gingivitis) Severe inflammation, marked redness and hypertrophy, ulceration, tendency to spontaneous bleeding (Severe Gingivitis) Bleeding on Probing (BOP) BOP tendency will be registered 20 seconds after probing. The following are the codes which will form the basis of the assessment for BOP (Lang, 1990) 0. Absent (on probing there is no bleeding)

1. Present (Bleeding after 20s of probing) Probing Depth (PD) The PD will be measured to the nearest millimeter on the scale of the periodontal probe (Badersten, 1990).WHO Probe (CPITN Probe): The tip of the probe has a 0.5 mm ball at the tip and millimeter marking at 3.5, 8.5 and 11.5 mm and the color coding are 3.5 to 5.5 mm.

Clinical Attachment Loss (CAL) It is measured by the distance between the cemento-enamel junction (CEJ) and the gingival margin (GM).

Following is the classification of CAL Slight = 1-2 mm, Moderate = 3-4 mm, Severe = ≥ 5mm). Pain associated with tooth movement To study the analgesic effect of Low- Level Laser Therapy, numerical rating scale (NRS) will be used.This scale ranges from 0 to 10 where 0 denotes no pain and 10 signify unbearable pain. NRS scale is valid, reliable and easier to be used by patients as compared to other similar scales like VAS (visual analogue scale).

A Performa to record the level of pain has been designed which will be given to all the patients after the application of force. Patients will be advised to record the pain intensity for 7 days, experienced 2 hours after force application to both groups experimental and controlled. Pain will be recorded by patients every 3 weeks when sequences wires are activated. Experimental and control groups will be compared to evaluate the effects of applied therapies on pain associated with tooth movement. The procedure will be the same for both groups to clarify the research question that whether the applied therapy with conventional brackets is more beneficial in terms of pain reduction or not?

Rate of tooth movement:

To study the effect of Low- Level Laser Therapy on tooth movement the study models to access tooth movement will be taken in all visits from 0 to 6th visit. The samples will be obtained from both groups consisted of Class I malocclusion with mild crowding patients treated orthodontic ally without extractions and patients with moderate irregularity scale of the index will be 2-4 according to Little's Irregularity Index (Little, 1975).

Dental cast measurements The T0 to T6 maxillary dental casts will be used. All dental cast measurements will be measured with a Laser scanner. 3D scanning of the models will be performed with HIROX 700 (Stereomicroscope) at USM Malaysia.

All will be in linear measurements, in millimeters, described as follows:

(A) Maxillary incisor irregularity. (B) Intercanine width (A; INTERC): The linear distance between the cusp tips of the maxillary canines. When there is a facet, the cusp tip will be estimated (Fig 2).

(C) Inter-premolar widths (INTERPB and INTERPB'): The linear distance between left and right central fossae of the maxillary first (B) and second (B') premolars (Fig 2).

(D) Intermolar width (C; INTERMOL): The linear distance between the mesiobuccal cusps tips of the maxillary first molars. When there is a facet, the cusp tip will be estimated .

(E) Arch length (D + E; LENGTH): The linear distance along the mid line from the interincisal midline to the mesial contact of the first molars .

(F) Arch perimeter (F; PERIM): The distance in millimeters from the mesial dental contact of the left first molars to the mesial dental contact of the right first molars.

Statistical analysis Statistical analyses and calculations will be performed with SPSS software version 22 (Chicago, USA). First, to assess the normality of data, investigatore will use the Shapiro-Wilk test. Investigators will use bifactorial variance (ANOVA) for analysis of repeated measurements (Lin, 2007).

P value less than 0.05 will be considered significant. Financial support and sponsorship Nil. Conflicts of interest There are no conflicts of interest.

ELIGIBILITY:
Inclusion Criteria:

1. Selected patients will be Pakistani ethnic background.
2. Age 18 to 30 years.
3. Patients with class 1 with mild crowding (severity of malocclusion) according to little irregularity index to avoid individual variations. (Little, 1975)
4. Patient with healthy periodontium with no any sign of gingival inflamation.
5. Patients who indicated for orthodontic treatment with fixed appliances started with the conventional ligated brackets.
6. Patients who will sign consent for participation in research and use of collected specimen/data for future reference.
7. Patients who are able to read and understand English language because consent forms available only in language of English.
8. Patients with ovoid arch form to compact with laser assisted tray.

Exclusion Criteria:

1. Patients on medications which alter the gingival health e.g. Phenytoin (Dilantin), Cyclosporine A (Sandimmun), Nifedipine (Adalat), Corticosteroids, contraceptive pills.
2. Patients on those medications which alter the bone metabolism or tooth movement e.g. NSAIDs, Corticosteroids, Bisphosphonates etc.
3. Patients with following disorder: Diabetes Type 1 and 2, Osteoporosis, Platelet disorders, Vitamin C deficiency, vascular conditions, Leukemia, HIV infection, crohn's disease.
4. Patients with pregnancy.
5. Patients with parafunctional habits, TMJ dysfunction, craniofacial malformation, multiple missing teeth, impacted teeth except third molars, or periodontally compromised patients will be excluded from the study.

   -

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Pain associated with tooth movement: numerical rating scale | A Performa to record the level of pain will be given to participants and advised to record the pain intensity for 7 days, experienced 2 hours after force application,as a primary outcome participants in experimental group may feel lesser pain.
  To study the analgesic effect of Low- Level Laser Therapy, numerical rating scale (NRS) will be used (Bertl, 2012). This scale ranges from 0 to 10 where 0 denotes no pain and 10 signify unbearable pain. NRS scale is valid, reliable and easier to be used by patients as compared to other similar scales like VAS (visual analogue scale) (Brunelli, 2010).

SECONDARY OUTCOMES:
Gingival index | To take examinations on each orthodontic treatment visit after every three weeks till six months of all participants of both groups,may show improvement in experimental group
  The examination was performed by using a blunt probe (Löe, 1963).Measurement Zero healthy condition and rating at 3 shows severity of disease Score Criteria 0.No inflammation
  1. Mild inflammation, slight change in color, slight edema, no bleeding on probing (Mild Gingivitis)
  2. Moderate inflammation, moderate glazing, redness, bleeding on probing (Moderate Gingivitis).
  3. Severe inflammation, marked redness and hypertrophy, ulceration, tendency to spontaneous bleeding (Severe Gingivitis)
Bleeding on Probing | To take examinations on each orthodontic treatment visit after every three weeks till six months
  BOP tendency will be registered 20 seconds after probing. The following are the codes which will form the basis of the assessment for BOP (Lang, 1990) 0. Absent (on probing there is no bleeding)
  1. Present (Bleeding after 20s of probing)
Clinical Attachment Loss | To take examinations on each orthodontic treatment visit after every three weeks till six months
  It is measured by the distance between the cemento-enamel junction (CEJ) and thegingival margin (GM). (Armitage, 2004) Following is the classification of CAL Slight = 1-2 mm, Moderate = 3-4 mm, Severe = ≥ 5mm)
Probing Depth | To take examinations on each orthodontic treatment visit after every three weeks till six months
  The PD will be measured to the nearest millimeter on the scale of the periodontal probe (Badersten, 1990). WHO Probe (CPITN Probe): The tip of the probe has a 0.5 mm ball at the tip and millimeter marking at 3.5, 8.5 and 11.5 mm and the color coding are 3.5 to 5.5 mm.
Rate of tooth movement: | To study the effect of Low- Level Laser Therapy on tooth movement the study models to access tooth movement will be taken in all visits from 0 to 6th visit.
  The impressions for study models for measurement of tooth movement will be obtained from both groups consisted of Class I malocclusion with mild crowding patients treated orthodontically without extractions and patients with moderate irregularity scale of the index will be 2-4 according to Little's Irregularity Index.

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan Hospital for Women Karimabad A secondary Hospital ofAga khan university Hospital, Karachi, Sindh Pakistan, Pakistan

IPD SHARING:
Plan to Share IPD: No
Still in the process of registration of study and ethical approval so want to share study on later stages

REFERENCES:
- [Result] Aihara N, Yamaguchi M, Kasai K. Low-energy irradiation stimulates formation of osteoclast-like cells via RANK expression in vitro. Lasers Med Sci. 2006 Apr;21(1):24-33. doi: 10.1007/s10103-005-0368-4. Epub 2006 Mar 28. PMID 16568210
- [Result] Hamdan AM. The relationship between patient, parent and clinician perceived need and normative orthodontic treatment need. Eur J Orthod. 2004 Jun;26(3):265-71. doi: 10.1093/ejo/26.3.265. PMID 15222710
- [Result] Jones ML, Chan C. Pain in the early stages of orthodontic treatment. J Clin Orthod. 1992 May;26(5):311-3. No abstract available. PMID 1430181
- [Result] Jones ML, Richmond S. Initial tooth movement: force application and pain--a relationship? Am J Orthod. 1985 Aug;88(2):111-6. doi: 10.1016/0002-9416(85)90234-9. PMID 3861096
- [Result] Lim HM, Lew KK, Tay DK. A clinical investigation of the efficacy of low level laser therapy in reducing orthodontic postadjustment pain. Am J Orthod Dentofacial Orthop. 1995 Dec;108(6):614-22. doi: 10.1016/s0889-5406(95)70007-2. PMID 7503039
- [Result] Qadri T, Miranda L, Tuner J, Gustafsson A. The short-term effects of low-level lasers as adjunct therapy in the treatment of periodontal inflammation. J Clin Periodontol. 2005 Jul;32(7):714-9. doi: 10.1111/j.1600-051X.2005.00749.x. PMID 15966876